CLINICAL TRIAL: NCT04357717
Title: Clinical Evaluation of ExoDx™ Prostate (IntelliScore) in Men With Prior Negative Prostate Biopsy Presenting for a Repeat Biopsy
Brief Title: ExoDx Prostate Evaluation in Prior Negative Prostate Biopsy Setting
Status: Terminated | Type: Observational
Why Stopped: project reprioritization
Sponsor: Exosome Diagnostics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ECT2018-001
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer
Keywords: exosome; ExoDx Prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: ExoDx Prostate — Urine-based biomarker tool to support decision to biopsy in patients with PSA between 2-10ng/ml

SUMMARY:
The study is designed to confirm the performance of the ExoDx Prostate test in prior negative biopsy patients now presenting for a repeat prostate biopsy.

Note: ExoDx Prostate test results are collected for correlation to biopsy results and are not disclosed to the physician or study subject.

DETAILED DESCRIPTION:
Primary Endpoint:

Evaluate the correlation of the ExoDx Prostate test results with the outcome of prostate biopsies in a prior negative repeat biopsy patient cohort.

Secondary Endpoints (exploratory):

1. Evaluate the clinical performance of the ExoDx Prostate test at the cut-point of 15.6 defined for the initial biopsy patient cohort.
2. Associate ExoDx Prostate test results with other ancillary studies including the use of radiographic imaging (e.g. multiparametric MRI).
3. Evaluate the correlation of ExoDx Prostate as a function of risk. It is known that a higher ExoDx Prostate score correlates to a higher risk of finding prostate cancer, including HGPC, upon biopsy.
4. Evaluate ExoDx Prostate with and without inclusion of standard of care parameters such as PSA, ethnicity, DRE, age and family history.

ELIGIBILITY:
Inclusion Criteria:

* 50+ years of age
* Clinical suspicion for prostate cancer
* Elevated Prostate-specific Antigen between 2.0-10 ng/ mL
* At least one (1) prior negative prostate biopsy

Exclusion Criteria:

* Use of medications or hormones that are known to affect serum PSA levels within 3-6 months of study enrollment including 5-alpha-reductase inhibitors used in the treatment of an enlarged prostate gland (benign prostatic hyperplasia). Drugs in this class are finasteride (Proscar, Propecia) and dutasteride (Avodart).
* Clinical symptoms of urinary tract infection (including prostatitis) at the time of enrollment.
* History of prostate cancer.
* History of invasive treatments for benign prostatic hypertrophy (BPH) or lower urinary track symptoms within 6 months of study enrollment.
* No known hepatitis status (all types) and/or HIV documented in patient's medical record.
* Patients with history of concurrent renal/bladder tumors.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Study Population: Men, aged 50yrs or older with an elevated PSA between 2-10ng/ml and at least one prior negative prostate biopsy
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2020-03-15 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Correlation of the ExoDx Prostate test results with the outcome of prostate biopsies in a prior negative repeat biopsy patient cohort. | 6 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chesapeake Urology Research Associates, Baltimore, Maryland
  - New Jersey Urology, Voorhees Township, New Jersey